CLINICAL TRIAL: NCT00899353
Title: Inhibition of Nuclear Factor Kappa B for Prevention of Disease Progression in Indolent B Cell Malignancies
Brief Title: Prevention of Disease Progression in Early Stage Indolent B Cell Malignancies. (SMM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original Principal Investigator left the institution.
Sponsor: Marshall University (Other)
Collaborators: Edwards Foundation, Inc. (Other)
Responsible Party: Principal Investigator, W. Elaine Hardman, Ph.D., W. Elaine Hardman, Ph.D., Marshall University School of Medicine, Professor of Biochemistry and Microbiology, Marshall University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MU9230
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Chronic Lymphocytic Leukemia
Keywords: ES-CLL; MGUS; SMM; Early Stage - Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega 3 supplement (Experimental): Omega 3 supplement will be added to diet, 3 capsules per day for one month then 6 capsules per day for one month then 9 capsules per day as tolerated
  Interventions: Dietary Supplement: Omega 3 Fatty Acid

INTERVENTIONS:
Dietary Supplement: Omega 3 Fatty Acid — Omega 3 supplementation will be initiated at three 1250 mg capsules daily for the first month. If dose is well tolerated, it will be increased to six 1250 mg capsules daily for 30 days, and finally to nine 1250 mg capsules daily. Treatment period is 12 months.
  Other Names: Res-Q® 1250

SUMMARY:
Escalating doses of Omega 3 Fatty Acids are being used in patients who have early stage Chronic Lymphocytic Leukemia (ES-CLL), Monoclonal Gammopathy of Undetermined Significance (MGUS), or Smoldering Multiple Myeloma (SMM), whose disease does not currently require treatment. The primary aim of the study is to determine if the Omega 3 supplementation will help prevent or delay progression of the disease to a stage that requires treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age.
* Must be free of other medical conditions that would decrease life expectancy to less that 12 months.
* Must be free of Omega 3 supplements or other fish oil containing nutritional supplements for a minimum of two months prior to enrollment.
* Must have a ECOG performance status of 0,1 or 2.

Exclusion Criteria:

* Any life-threatening condition such as (but not limited to) advanced heart disease, kidney or liver failure with an expected survival of less than 12 months.
* Any other active malignancy.
* Women who are pregnant or lactating.
* Individuals unable to give informed consent.
* Individuals with known allergy or intolerance to fish oil supplements.
* Any patient with an active bleeding diatheses or disorder.
* ECOG performance status of 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanda E Hardman, Ph.D., Principal Investigator — Professor Marshall University School of Medicine
Locations (1):
- Edwards Comprehensive Cancer Center, Huntington, West Virginia, United States

REFERENCES:
- [Derived] Witte TR, Salazar AJ, Ballester OF, Hardman WE. RBC and WBC fatty acid composition following consumption of an omega 3 supplement: lessons for future clinical trials. Lipids Health Dis. 2010 Mar 22;9:31. doi: 10.1186/1476-511X-9-31. PMID 20307284

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega 3 Supplementation: Baseline blood specimens were obtained. All participants were then assigned to consume three, 1250mg omega 3 supplement capsules per day (providing 2.4g of omega 3 total) for one month, the first period. Blood was obtained and participants were assigned to consume six, 1250mg capsules of omega 3 per day (providing 4.8g of omega 3)for one month, the second period. Blood was again obtained and participants were assigned to consume 9 capsules of omega 3 per day, providing 7.2g of omega 3,the third period.
Period: Overall Study
Arm/Group | Omega 3 Supplementation
Started | 16
Completed | 11
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Omega 3 Supplementation
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Activated Nuclear Factor Kappa B (NFkB) in Peripheral Blood Lymphocytes From Patients With Early Stage Chronic Lymphocytic Leukemia (CLL) Before, During and After Consumption of an Omega 3 Supplement.
Description: Peripheral lymphocytes were isolated from the blood using Ficoll-Paque gradient. Nuclear Factor Kappa B activation was analyzed using Thermo Scientific Transcription Factor kit for NFkB p50, according to manufacturer's protocol. Protein extracts containing 1-15µg of protein/well were added in triplicates. Luminescence resulting from a reaction with bound NFkB was detected using a Berthold Centro LB960 Luminometer and analyzed with MikroWin 2000 ver. 1.08. NFkB activity was normalized by luminescence units/µg of protein per well.
Time Frame: baseline, and post supplement month 1(3 capsules/day), month 2 (6capsules/day), month 3 (9 capusules/day), month 6 (9 capusules/day), month 9 (9 capusules/day), month 12 (post supplement)
Population: NFkB activation of all patients diagnosed with early stage CLL at baseline and following omega 3 consumption. Patients are further separated into high (> median, n=7) and low initial baseline (< median, n=6) NFkB. Patients included must have had one baseline and at least one period of omega 3 consumption. Not all patients completed all periods
Measure: Mean (Standard Error); unit: 10^6 NFkB Luminescence units/µg protein
Groups:
- Baseline Nuclear Factor Kappa B Activation: Baseline nuclear factor Kappa B (NFkB) activation in isolated lymphocytes from patients with early stage chronic lymphocytic leukemia.
- Nuclear Factor Kappa B Activation Following 3 Capsules Per Day: Nuclear factor Kappa B (NFkB)activation in isolated lymphocytes from patients with early stage chronic lymphocytic leukemia following consumption of 3 capsules per day (2.4 g of omega 3 per day). Each 1250mg capsule provided 800mg of omega 3.
- Nuclear Factor Kappa B Activation Following 6 Capsules Per Day: Nuclear factor Kappa B (NFkB)activation in isolated lymphocytes from patients with early stage chronic lymphocytic leukemia following consumption of 6 capsules per day (4.8 g of omega 3 per day).Each 1250mg capsule provided 800mg of omega 3.
- Nuclear Factor Kappa B Activation Following 9 Capsules Per Day: Nuclear factor Kappa B (NFkB)activation in isolated lymphocytes from patients with early stage chronic lymphocytic leukemia following consumption of 9 capsules per day (7.2 g of omega 3 per day). Each 1250mg capsule provided 800mg of omega 3.
- Nuclear Factor Kappa B Activation Post Supplement: Nuclear factor Kappa B (NFkB)activation in isolated lymphocytes from patients with early stage chronic lymphocytic leukemia following discontinued consumption of omega 3.
Arm/Group | Baseline Nuclear Factor Kappa B Activation | Nuclear Factor Kappa B Activation Following 3 Capsules Per Day | Nuclear Factor Kappa B Activation Following 6 Capsules Per Day | Nuclear Factor Kappa B Activation Following 9 Capsules Per Day | Nuclear Factor Kappa B Activation Post Supplement
Number analyzed (Participants) | 15 | 12 | 12 | 10 | 8
10^6 NFkB Luminescence units/µg protein
  Total Population | 7.2 (2.25) [0.945 to 231] | 4.1 (1.53) | 4.2 (1.15) | 0.7 (0.94) | 1.5 (0.86)
  Higher Initial Expressers | 12.8 (2.77) | 7.4 (2.41) | 6.4 (1.42) | 0.8 (0.20) | 1.6 (1.44)
  Lower Initial Expressers | 0.8 (0.27) | 0.9 (0.37) | 1.5 (0.80) | 0.6 (0.11) | 1.3 (1.16)
Statistical Analysis 1: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 3 Capsules Per Day; Omnibus analysis. Statistical significance was determined by Games Howell Multiple Comparison test. Significance was determined as α< 0.05. Analysis based on global response; Test type: Superiority or Other; p = 0.78, ANOVA; Games-Howell Correction was applied to adjust for unequal variances, unequal sample size and for non-parametric distribution; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-5.0 to 11.2], Standard Error of Mean 2.7
Statistical Analysis 2: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 6 Capsules Per Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.75, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-4.6 to 10.7], Standard Error of Mean 2.5
Statistical Analysis 3: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 9 Capsules Per Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.08, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.6, 95% CI 2-sided [-0.6 to 13.7], Standard Error of Mean 2.3
Statistical Analysis 4: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Post Supplement; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.17, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-1.6 to 13.2], Standard Error of Mean 2.4
Statistical Analysis 5: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 3 Capsules Per Day; Omnibus analysis. Statistical significance was determined by Games Howell Multiple Comparison test. Significance was determined as α< 0.05. Analysis based on High Initial NFkB Activation Expressers; Test type: Superiority or Other; p = 0.61, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-6.5 to 17.2], Standard Error of Mean 3.7
Statistical Analysis 6: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 6 Capsules Per Day; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.32, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [-4.1 to 16.8], Standard Error of Mean 3.1
Statistical Analysis 7: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 9 Capsules Per Day; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.03, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.0, 95% CI 2-sided [1.6 to 22.3], Standard Error of Mean 2.8
Statistical Analysis 8: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Post Supplement; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.04, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.1, 95% CI 2-sided [0.5 to 21.8], Standard Error of Mean 3.1
Statistical Analysis 9: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 3 Capsules Per Day; Omnibus analysis. Statistical significance was determined by Games Howell Multiple Comparison test. Significance was determined as α< 0.05. Analysis based on Low Initial NFkB Activation Expressers; Test type: Superiority or Other; p = 1.00, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.5 to 1.2], Standard Error of Mean 0.4
Statistical Analysis 10: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 6 Capsules Per Day; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.88, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-3.5 to 2.3], Standard Error of Mean 0.7
Statistical Analysis 11: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Following 9 Capsules Per Day; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.98, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0], Standard Error of Mean 0.3
Statistical Analysis 12: Comparison: Baseline Nuclear Factor Kappa B Activation vs Nuclear Factor Kappa B Activation Post Supplement; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.98, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-6.6 to 5.3], Standard Error of Mean 1.2

2. Primary Outcome: The Degree of Change in Tumor Mass Measurements During and After Omega-3 Supplementation as Evaluated by Standard Clinical Tests of Disease Activity.
Description: Patients diagnosed with early stage (asymptomatic) CLL were supplemented with escalating doses of omega-3 (n-3) fatty acids (2.4 g of n-3/day up to 7.2 g of n-3/day). Given that these patients are asymptomatic and did not require treatment, measures of tumor mass during and after omega-3 supplementation, as evaluated by standard clinical tests of disease activity, were not performed. Instead, absolute lymphocyte counts (ALC), as a measure of tumor burden, was evaluated before and after omega-3 supplementation. Data represents the fold change in ALC post omega-3 consumption as compared to baseline ALC.
  Patients with MGUS or SMM were not enrolled into this study.
Time Frame: Baseline, month 1, month 2, month 3, month 6, month 9, 12 months
Population: Patients who's absolute lymphocyte counts were known prior to omega-3 initiation (baseline) and after omega-3 consumption were included in this analysis. Patients who's ALC was unknown prior to omega-3 initiation or after omega-3 consumption were excluded.
Measure: Number; unit: Fold Change
Groups:
- Fold Change in ALC-Patient 1; Fold Change in ALC-Patient 2; Fold Change in ALC-Patient 3; Fold Change in ALC-Patient 4; Fold Change in ALC-Patient 5; Fold Change in ALC-Patient 6; Fold Change in ALC-Patient 7; Fold Change in ALC-Patient 8; Fold Change in ALC-Patient 9; Fold Change in ALC-Patient 10; Fold Change in ALC-Patient 11; Fold Change in ALC-Patient 13; Fold Change in ALC-Patient 14: Fold change in ALC after omega-3 consumption as compared to baseline ALC.
Arm/Group | Fold Change in ALC-Patient 1 | Fold Change in ALC-Patient 2 | Fold Change in ALC-Patient 3 | Fold Change in ALC-Patient 4 | Fold Change in ALC-Patient 5 | Fold Change in ALC-Patient 6 | Fold Change in ALC-Patient 7 | Fold Change in ALC-Patient 8 | Fold Change in ALC-Patient 9 | Fold Change in ALC-Patient 10 | Fold Change in ALC-Patient 11 | Fold Change in ALC-Patient 13 | Fold Change in ALC-Patient 14
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Fold Change | 1.62 | 1.71 | 0.78 | 0.96 | 1.32 | 1.08 | 1.00 | 0.92 | 1.49 | 1.05 | 1.16 | 1.03 | 1.22

ADVERSE EVENTS:
Groups:
- Adverse Effects: Serious adverse effects associated with omega 3 fatty acid consumption.
Arm/Group | Adverse Effects
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Effects (N=16)
Diarrhea (Gastrointestinal disorders) | 4 (5) — Grade 1 and 2 Diarrhea in participants consuming 6 or 9 capsules per day (4.8 or 7.2g per day)
Nausea (General disorders) | 2 (3) — Participants were consuming 6 or 9 capsules per day (4.8 or 7.2g per day)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes